CLINICAL TRIAL: NCT05373069
Title: BENEFIT OF MECHANICAL ISCHEMIC PRECONDITIONING ON TOLERANCE OF ADIPOSE TISSUE TO ISCHEMIA REPERFUSION OF TYPE DIEP (DEEP INFERIOR EPIGASTRIC PERFORATOR) FREE FLAPS.
Acronym: PRIMIDIEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: INSERM Bichat hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP201173; 2021-A00173-38 (Other: ANSM)
Record Dates: First submitted 2022-03-04; First posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer
Keywords: Breast reconstruction; Ischaemic preconditioning; DIEP flap
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group intervention (Experimental): PIM - DIEP
  Interventions: Procedure: Mechanical ischemic preconditioning of diep-type flap

INTERVENTIONS:
Procedure: Mechanical ischemic preconditioning of diep-type flap — Mechanical ischemic preconditioning: Performing series of reperfusion ischemia on the flap pedicle, before cold ischemia of the flap (flap harvesting before vascular mechanical anastomoses at the recipient site)
  * 10 min of clamping with single-use microvascular forceps
  * 10 min declamping
  * 10 min of tightening with pliers
  * 10 min declamping Either preconditioning for 40 minutes, simulating 2 cycles of ischemia reperfusion prior to flap harvesting and cold ischemia before revascularization.

SUMMARY:
Breast cancer is the most common cancer amongst women in terms of frequency, with more than 50 000 newly diagnosed cases per year in France. The average 5-year survival rate for women with breast cancer is around 85%. Surgical treatment by total mastectomy concerns around 30% of cases. For patients who have been treated for breast cancer by total mastectomy, secondary breast reconstructions are often carried out via excess abdominal fat flaps of DIEP type.

Postoperative partial fat necrosis is a common complication of breast reconstruction. This necrosis is qualified as pathological when it is palpable or when there are symptoms leading to pain, deformation, or leakage. Necrosis occurs in the first 6 months after surgery. Diagnosis is carried out by the detection of a nodule of fat necrosis measuring at least 5 mm on the ultrasound.

Partial flat necrosis results from ischemia reperfusion (IR) to the fat tissues during reconstruction. IR leads to inflammatory lesions, edema, capillary occlusion that can lead to tissue necrosis. The deleterious impact of IR has been shown on the organs (liver, kidney) on muscular, cutaneous and adipose tissues in humans and animals.

Ischaemic preconditioning is a procedure used in organ transplant surgery, allowing a better tolerance of the graft for ischemia reperfusion, without further complications. It is used in usual practice for kidney or liver transplants; short cycles of ischemia reperfusion are carried out on the organ pedicle before harvesting using cold ischemia (out of the donor's body) pre-transplant.

Ischaemic preconditioning before reconstruction has been studied in animal models but not in human reconstruction surgery, although it seems to be beneficial. For patients undergoing total mastectomy after being diagnosed with breast cancer, we hypothesize that ischaemic preconditioning, usually used for organ transplants, could decrease adipose tissue lesions caused by ischemia reperfusion after breast reconstruction with DIEP (deep inferior epigastric perforator) flaps.

DETAILED DESCRIPTION:
This is a phase 2 monocentric study, following the 2 step Simon Minimax design.

We will be carrying out cycles of ischemic preconditioning for 40 minutes, simulating 2 cycles of ischemia-reperfusion (per 10min) prior to flap harvesting and cold ischemia before revascularization.

The pre operation visit will occur between M3 and M1 before the scheduled operation date. The visit will be carried out by the surgeon who will inform the patient of the study.

The inclusion visit (D0) will be carried out by the investigator the day before surgery (collection of signed consent form). The surgery will be carried out as usual: breast reconstruction with DIEP type flap. Modification of the intervention for the study: preconditioning of the flap (for patients) and 3 biopsies.

During post-operative hospitalization, usual visits will be carried out twice a day (not specifically for the study) by an doctor (to check for vascular damage, hematoma, infection, cutaneous necrosis, leakage and scar separation).

After postoperative discharge, 4 follow up visits are planned which correspond to 3 postoperative consultations at the hospital (to check for vascular damage, hematoma, infection, cutaneous necrosis, leakage and scar separation) at D21 (+/- 2 days), M1 (+/- 2 days), M3 (+/- 15 days, same assessment plus search for palpable, painful or deforming nodules) and M6 (+/- 15 days, last visit) plus a mammary ultrasound (this is the only supplementary assessment carried out for the study, Tenon hospital).

ELIGIBILITY:
Inclusion Criteria:

* female with age ≥ 18
* Secondary unilateral breast reconstruction using DIEP
* Signed consent form
* Beneficiary of a social security scheme

Exclusion Criteria:

* Smoking: active or quit since < 2 months, contraindication for flap surgery
* Pregnancy: contraindication for surgery
* Immediate breast reconstruction, at the same time as the mastectomy (increases cutaneous complications and different surgical technique)
* Bilateral breast reconstruction (increases operation time and post operation complications)
* Patient under curatorship or guardianship
* Patient deprived of their liberty, and patient undergoing psychiatric care
* Risk factor for DIEP complication such as: previous surgical procedures performed on the abdomen, carcinological treatments and severe comorbidities of the patient.
* Risk factors for complications of mechanical preconditioning. Soft tissue inflammation or osteomyelitis, peripheral arterial occlusive disease, vasculitis,
* Participation in another interventional study
* Any contraindication to general anesthesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Number of successes of the technique defined by the absence of pathological postoperative fat necrosis | 6 months post operation
  Number of successes of the technique defined by the absence of pathological postoperative fat necrosis to evaluate the efficacy of ischaemic preconditioning on the tolerance of the adipose tissue to the ischemia-reperfusion of DIEP flaps

SECONDARY OUTCOMES:
to evaluate the efficacy of ischaemic preconditioning on the tolerance of the skin (cutaneous necrosis, scar separation) to the ischemia-reperfusion of DIEP flaps | 6 months post operation
  proportion of patients with skin necrosis
Presence of skin necrosis within 6 months postoperatively defined by (occurrence of one or more of the three subcited elements | 6 months post operation
  * Skin infection
  * Skin necrosis of the flap
  * Scar disunion
Proportion of overall reconstruction failures: postoperative flap loss at M6: flap removal for total necrosis | 6 months post operation
Rate of subclinical cystosteatonecrosis (detected by ultrasound at M6: presence of one or more nodules, measuring more than 5mm but having no clinical repercussions) | 6 months post operation
to evaluate the proportion of overall failure after DIEP type flaps. | 6 months post operation
  Proportion of overall reconstruction failure (need to remove the flap for total necrosis)
to evaluate the proportion of subclinical cytosteatonecrosis | 6 months post operation
  rate of subclinical cysteatonecrosis

CONTACTS AND LOCATIONS:
Overall Officials: Sarra CRISTOFARI, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service Plastique, Reconstruction, Esthétique, Hôpital TENON- APHP, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided